CLINICAL TRIAL: NCT07018414
Title: The Effect of Abdominal Massage on Gastric Residual Volume and Abdominal Distension in Surgical Intensive Care Patients: A Randomized Controlled Trial
Brief Title: Abdominal Massage for Gastric Residual Volume in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ABMGRVSICU
Record Dates: First submitted 2025-05-23; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gastric Residual Volume; Abdominal Distension; Enteral Nutrition; Massage Therapy
Keywords: Enteral Nutrition; Gastric Emptying; Abdominal Distension; Intensive Care Units, Surgical; Postoperative Care; Gastrointestinal Motility Disorders; Critical Illness; Massage Therapy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: This study utilized a parallel assignment model, in which participants were randomly assigned to either the intervention group (receiving abdominal massage) or the control group (receiving standard care) in a 1:1 ratio. Each participant received only one type of intervention throughout the study period. The intervention was applied twice daily for 20 minutes over three consecutive days.
Masking Description: This study was conducted as an open-label trial, with no masking of participants, healthcare providers, or outcome assessors. Due to the nature of the intervention (abdominal massage), blinding was not feasible. However, data collection and statistical analyses were performed by researchers not involved in delivering the intervention to minimize potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage Group (Experimental): Patients in this group received abdominal massage for 20 minutes, twice daily, for three consecutive days after the initiation of enteral nutrition.
  Interventions: Behavioral: Abdominal Massage
- Control Group (No Intervention): Patients in this group received standard postoperative care without abdominal massage.

INTERVENTIONS:
Behavioral: Abdominal Massage — Non-pharmacological intervention involving manual massage of the abdomen to support gastric motility and reduce gastric residual volume and abdominal distension in enterally fed surgical ICU patients.
  Arms: Abdominal Massage Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effect of abdominal massage on gastric residual volume (GRV) and abdominal distension in surgical intensive care patients receiving enteral nutrition. The intervention group received 20-minute abdominal massage sessions twice daily for 3 consecutive days. Outcomes included changes in GRV, abdominal circumference, feeding volume, and gastrointestinal tolerance parameters.

DETAILED DESCRIPTION:
Gastric residual volume (GRV) monitoring is commonly used in critically ill patients receiving enteral nutrition to assess gastrointestinal dysfunction, although current guidelines present conflicting recommendations regarding its necessity. Abdominal distension is a frequent complication during enteral feeding in surgical ICU patients. Non-pharmacological interventions such as abdominal massage have shown promise in improving gastrointestinal motility and enteral tolerance.

This study included 84 surgical ICU patients who met the inclusion criteria and were randomly assigned to intervention (n=42) and control (n=42) groups. The intervention group received abdominal massage twice daily for 20 minutes over three days. Data were collected using standardized forms and analyzed with appropriate statistical tests including independent samples t-test, Mann-Whitney U, repeated measures ANOVA, and chi-square tests. The findings suggest that abdominal massage may help stabilize GRV levels, reduce abdominal circumference, and increase nutritional intake without increasing complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Receiving enteral nutrition via nasogastric tube
* No prior abdominal surgery
* No invasive devices (e.g., drains, catheters) in the abdominal area

Exclusion Criteria:

* Receiving enteral nutrition via PEG or PEJ
* Receiving only parenteral nutrition
* History of abdominal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Amount of gastric residual volume (mL) | Day 3
  Starting from the first day of enteral nutrition, gastric residual volume (mL) will be recorded at regular intervals every day for 3 days. The amount of GRV changing from the first day to the 3rd day will be measured and analysed.
Change in abdominal circumference | Day 3
  Abdominal circumference will be measured on the first day of enteral feeding and abdominal circumference will be measured every day at the same time for 3 days. The change in abdominal circumference (cm) from baseline to Day 3 will be recorded.

SECONDARY OUTCOMES:
Amount of enteral feeding (mL/day) | Day 3
  The total amount of nutritional product taken on the first day of enteral nutrition will be recorded for 3 days. The amount taken from the beginning to the 3rd day will be recorded in ml/day.
Assessment of abdominal distension | Day 3
  On the first day of enteral nutrition, abdominal circumference will be measured and abdominal distension will be evaluated by auscultating bowel sounds and daily X-rays. The presence or absence of abdominal distension from the beginning to the 3rd day will be recorded.
Interruption of enteral nutrition | Day 3
  From the first day of starting enteral nutrition, the reasons for which continuous nutrition is interrupted (for example, going to another unit for radiological examination or re-operation for revision purposes, etc.) will be monitored and recorded for 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Seyrantepe Hamidiye Etfal Training and Research Hospital, Surgical Intensive Care Units, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data due to privacy concerns and institutional policy.